CLINICAL TRIAL: NCT05041452
Title: Multiparametric Cardio-hepatic MRI in Patients With Noncirrhotic Portal Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Julian Alexander Luetkens, Principal Investigator, Senior Physician, University Hospital, Bonn
Other Study IDs: 282/18
Record Dates: First submitted 2021-08-27; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Hypertension, Portal; Cardiomyopathies
Keywords: Cardiac MRI; Hepatic MRI
MeSH Terms: conditions — Hypertension, Portal; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Noncirrhotic portal hypertension (NCPH): Patients with non-cirrhotic portal hypertension (NCPH) with pre-sinusoidal (e.g., porto-sinusoidal vascular disease, portal vein obstruction, congenital hepatic fibrosis, biliary diseases,), sinusoidal (e.g., sinusoidal destruction in the setting of acute hepatic injury, inflammatory or toxic fibrosis, non-alcoholic steatohepatitis), or post-sinusoidal causes (Budd-Chiari syndrome, sinusoidal obstruction syndrome).
  Interventions: Diagnostic Test: Cardiac magnetic resonance scan
- Cirrhotic portal hypertension: Patients with cirrhosis and portal hypertension.
  Interventions: Diagnostic Test: Cardiac magnetic resonance scan

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance scan — Multiparametric cardiac magnetic resonance, including functional and structural parameters

SUMMARY:
The aim of this study is to use multiparametric MRI to investigate any differences in myocardial structure and function in patients with noncirrhotic portal hypertension compared with a control group with liver cirrhosis.

DETAILED DESCRIPTION:
The term "cirrhotic cardiomyopathy" (CCM) was defined in 2005 according to expert consensus at the "World Congress of Gastroenterology" in Montreal as a clinical phenotype in patients with liver cirrhosis consisting of systolic and diastolic dysfunction and a complementary criterion, such as electrophysiological changes, without the presence of a known underlying cardiac disease. For a long time, CCM was considered to result from toxic effects of alcohol consumption. The current view is that CCM is a separate entity independent of the various etiologies of liver cirrhosis. Thus, generally impaired liver function and portal hypertension with splanchnic vasodilation leads to altered hemodynamic conditions with central hypovolemia, increased activation of volume and baroreceptors, especially of the sympathetic nervous system, resulting in a "hyperdynamic syndrome" with increased cardiac stress. However, the contribution of portal hypertension to CCM is unclear.

With new MRI techniques such as cardiac T1 and T2 mapping and extracellular volume fraction (ECV), quantitative parameters are available to detect pathologies of the myocardium before they become detectable with conventional techniques in cardiac MRI or echocardiography.

The aim of this study is to use multiparametric MRI to investigate any differences in myocardial structure and function in patients with noncirrhotic portal hypertension compared with a control group with liver cirrhosis and to investigate a quantifiable correlation between cardiac, hepatic, and splenic parameters.

ELIGIBILITY:
Inclusion criteria:

1. noncirrhotic portal hypertension
2. age at least 18 years

Exclusion criteria:

1. underlying cardiac disease, e.g., coronary heart disease/myocardial infarction, myocarditis, cardiomyopathies of other causes, congenital heart disease
2. patients who are using a intrauterinpessare for contraception
3. pregnant and breastfeeding women
4. patients with contraindications for MRI (not suitebale metallic implants)
5. patients with contraindications for MRI contrast agents (renal insufficiency, allergy)

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with clinically diagnosed noncirrhotic portal hypertension who are being treated at the Medical Clinic and Polyclinic I of the University Hospital Bonn are included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-04-29 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial T1 relaxation time | Measurement will be performed within 2 weeks after MRI scan.
  T1 relaxation times will be obtained to asses acute myocardial injury and fibrosis. T1 maps will be analyzed using a segmental approach by region of interest analysis. T1 relaxation times are given in [ms].

SECONDARY OUTCOMES:
Myocardial T2 relaxation time | Measurement will be performed within 2 weeks after MRI scan.
  T2 relaxation times will be obtained to asses myocardial edema. T2 maps will be analyzed using a segmental approach by region of interest analysis. T2 relaxation times are given in [ms].
Myocardial ECV | Measurement will be performed within 2 weeks after MRI scan.
  Myocardial extracellular volume will be obtained to asses extracellular space/myocardial fibrosis. ECV values will be calculated using a segmental approach by region of interest analysis of native and contrast-enhanced T1 relaxation maps. ECV values are given in [%].
Myocardial strain | Measurement will be performed within 2 weeks after MRI scan.
  Cardiac magnetic resonance feature-tracking will be used to asses left ventricular longitudinal, circumferential and radial strain.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Bonn, Clinic for Diagnostic and Interventional Radiology, Bonn, North Rhine-Westphalia
  - University Hospital Bonn, Medical Clinic and Polyclinic I, Bonn, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No